CLINICAL TRIAL: NCT02365688
Title: Correlation of Multiple Invasive and Non-Invasive Hemodynamic Monitored Modalities to Support Goal Directed Fluid Therapy During Open Abdominal Surgery
Brief Title: Hemodynamic Response During Goal Directed Fluid Therapy in the OR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of consistent reference devices
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COVMOPR0436
Record Dates: First submitted 2014-09-09; First posted 2015-02-19 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Hemodynamic Instability
Keywords: Open Abdominal Surgical Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Initial bolus pre-incision (Other): Initial pre-incision bolus of 500 cc of fluids with hemodynamic response recorded
  Interventions: Procedure: Initial bolus pre-incision

INTERVENTIONS:
Procedure: Initial bolus pre-incision — Measured hemodynamic response to pre-incision bolus

SUMMARY:
The purpose of this study is to retrospectively evaluate the hemodynamic response to goal directed fluid therapy fluid during open abdominal surgery where goal directed fluid therapy is a standard of care after establishing a pre-incision baseline response to fluids.

DETAILED DESCRIPTION:
Electronic and annotated observation data to support an algorithm library

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years booked for an open abdominal procedure
2. American Society of Anaesthesiologists (ASA) Physical Status 1 - 3
3. Expected duration of surgical procedure to be ≥ 2 hours
4. Standard of care monitoring to include cardiac output

Exclusion Criteria:

1. Open chest surgical procedure expected
2. Cardiac arrhythmia such as atrial fibrillation.
3. Right Ventricular Failure
4. Aortic regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E Miller, MB ChB, FRCA, Principal Investigator — DUHS Department of Anestheiology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for new algorithm development

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients meeting the inclusion and exclusion criteria were recruited in the pre-op clinic. Recruitment started on 15-AUG-2014 with ended in January 2015.
Period: Overall Study
Arm/Group | Initial Bolus Pre-incision
Started | 18 (All subjects received a bolus of 500cc before first incision)
Completed | 18 (All subjects consented to an change in standard infusion volume pre-incision)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Self hemodynamic baseline before surgical incision.
Arm/Group | Initial Bolus Pre-incision
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 58 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Hemodynamic Response to Fluid Resuscitation
Description: Physiological parameters compared before and after fluid bolus for fluid resuscitation.
Time Frame: Up to 6 hours but not to exceed duration of surgical procedure
Population: Reference devices were in disagreement so the algorithm could not be verified
Arm/Group | Initial Bolus Pre-incision
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Two weeks. Consent in pre-op clinic to end of surgical procedure
Groups:
- Pre-surgical Bolus: Pre-surgical bolus of 500 cc before incision rather than during incision for baseline hemodynamic data
Arm/Group | Pre-surgical Bolus
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-surgical Bolus (N=18)
Hypertension (Surgical and medical procedures) | 1 (1) — Hypertensive event during open abdominal procedure
Blood Loss (Surgical and medical procedures) | 1 (1) — Excessive blood loss during the open abdominal procedure managed by fluid resuscitation

LIMITATIONS AND CAVEATS:
Reference devices did not agree so trial terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No